CLINICAL TRIAL: NCT00828022
Title: A Single-Institution, Open-Label, Single-Arm phase1/2 Study of Measles Vaccine as Consolidation in Patients With Measles Virus-Positive, Stage 3B/4 Non-Small Cell Lung Cancer
Brief Title: Measles Vaccine in Patients With Measles Virus-Positive, Advanced Non-Small Cell Lung Cancer
Acronym: SMC4692
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Prof. Samuel Ariad, Department of Oncology, Soroka Medical Center, Beer Sheva
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sor469208ctil
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Non-Small Cell Lung Cancer; Measles
Keywords: measles-positive NSCLC; measles vaccine; consolidation; Stage 3B with pleural effusion or stage 4 non-small cell lung cancer in remission
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Measles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: attenuated measles vaccine — 4-week apart, two vaccines starting 4 weeks after last chemotherapy

SUMMARY:
The objectives of the study are to assess the efficacy and safety of live, attenuated measles vaccine as consolidation therapy in patients with measles-positive, non-small cell lung cancer with locally-advanced (stage 3B with pleural effusion) or metastatic (stage 4) tumors in remission.

DETAILED DESCRIPTION:
This is a single-institution, non-randomized phase 1/2 study in patients with locally-advanced or metastatic NSCLC in remission after receiving standard systemic chemotherapy of four cycles of combination chemotherapy consisting of four cycles of cisplatin combined with vinorelbine.

ELIGIBILITY:
Inclusion Criteria:

* Patients in remission after first-line chemotherapy

Exclusion Criteria:

* Progressive disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-03

PRIMARY OUTCOMES:
To assess progression-free survival (PFS) and overall survival (OS) in patients with NSCLC in remission receiving subcutaneous live-attenuated measles virus vaccine as consolidation therapy in patients with measles-positive tumors. | 2-years

SECONDARY OUTCOMES:
To evaluate additional measures of efficacy, safety, and disease/treatment-related symptoms. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Soroka Medical Center, Beersheba, Israel